CLINICAL TRIAL: NCT03392623
Title: DNA Methylation in Malar Melasma and Its Change by Sunscreen, Retinoic Acid and Niacinamide.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo-Cazares, Medical Doctor, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 71-15
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Melasma
Keywords: Epigenetics, Malar melasma,
MeSH Terms: conditions — Melanosis | interventions — Tretinoin; Niacinamide; Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double bind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Control group (Other): Macules of melasma without any treatment
  Interventions: Device: colorimetry measurement
- Niacinamide group (Experimental): Macules of melasma treated with topical Niacinamide cream 4% for 8 weeks
  Interventions: Device: colorimetry measurement; Drug: Niacinamide
- Retinoic acid group (Experimental): Macules of melasma treated with topical retinoic acid 0.05% for 8 weeks
  Interventions: Drug: Retinoic acid; Device: colorimetry measurement
- Sunscreen group (Placebo Comparator): Macules of melasma treated with sunscreen cream with a 50 sun protection factor for 8 weeks
  Interventions: Device: colorimetry measurement; Drug: sunscreen

INTERVENTIONS:
Drug: Retinoic acid — topical administration in melasma lesions
  Other Names: Niacinamide; Sunscreen
  Arms: Retinoic acid group
Device: colorimetry measurement — Measurement of erythema and luminosity through a colorimeter
Drug: sunscreen — topical administration in melasma lesions
  Arms: Sunscreen group
Drug: Niacinamide — topical administration in melasma lesions
  Arms: Niacinamide group

SUMMARY:
BACKGROUND: Malar melasma has a chronic and recurrent character that may be related with epigenetic changes.

DETAILED DESCRIPTION:
OBJECTIVE: Recognize the DNA methylation status of the malar melasma and perilesional skin, and its change after treatment with 50 SPF sunscreen (S), 4% niacinamide (N), or 0.025% retinoic acid (RA). METHODS: Fifty-six lesion of 28 female patients without treatment were clinically evaluated, as also the expression of DNA methyl transferases 1 and 3 by real time-PCR (polymerase chain reaction amplification), immunohistochemistry and immunofluorescence. It was initially quantified and after 8 weeks of treatment with S, RA and N. RESULTS: Relative expression of DNA methyl transferases were significantly elevated compared with unaffected skin in all subjects indicating hypermethylation of DNA. Hypermethylation decreased by S (7 vs 3 times relative expression, p<0.05), RA (7 vs 2 times relative expression p<0.05), and N (7 vs 1 relative expression p<0.01) correlated with clinical improvement, this was also supported by immunohistochemistry and immunofluorescence. CONCLUSIONS: The investigators found hypermethylation of DNA in melasma lesions. Environmental factors such as sun radiation may induce DNA hypermethylation triggering hyperpigmentation trough the activation of pathways regulated by epigenetic modifications. Thus, decreasing methylation by sunscreen protection and the genetic transcription modification through N and RA, may allow their clinical improvement regardless its depigmenting effect.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of malar melasma by a specialist. No previous treatment at the beginning of the study.

Exclusion Criteria:

Use of medications associated with the development of melasma. Pregnant or lactating patients. Presence of concomitant diseases associated with the development of melasma. or other facial hyperpigmentations (thyroid, liver).

Have received treatment in the last 2 months. Regular use of sunscreen.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
improve in the level of DNA methylated | 8 weeks
  Decrease in levels of expression of DNA methyl transferases

SECONDARY OUTCOMES:
improve in the clinical severity of melasma | 8 weeks
  decrease in the MASI score

IPD SHARING:
Plan to Share IPD: No